CLINICAL TRIAL: NCT04670627
Title: Investigation of Molecular Biomarkers Associated With Occurrence of Seasonal Allergic Rhinitis (AR) In and Out of Active Allergy Season
Brief Title: Biomarkers in Nasal Samples of Seasonal Allergic Rhinitics
Acronym: GSK AR ELF
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-2258
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-07

CONDITIONS: Seasonal Allergic Rhinitis; Rhinovirus
Keywords: Seasonal Allergies
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Seasonal Allergic Rhinitics: Non-smoking males and females aged 18-70 years, inclusive with history of Seasonal Allergic Rhinitis defined by:
  Sensitization to at least one seasonal aeroallergen via skin prick testing (wheal =3 mm than negative control), AND History of physician-diagnosed seasonal allergic rhinitis, OR Symptoms consistent with seasonal allergic rhinitis, such as runny nose, nasal congestion, sneezing, or nasal pruritis.
- Control: Non-smoking males and females aged 18-70 years, inclusive with no history of physician-diagnosed allergic rhinitis and no history of seasonal runny nose, nasal congestion, sneezing or nasal pruritis. Negative results to a panel of aeroallergens via skin prick testing.

SUMMARY:
The purpose of this study is to analyze nasal samples for the presence of biomarkers of allergic inflammation as well as cold and flu infections, and compare these samples both in and out of an individual's active allergy season. 40 subjects who suffer from seasonal allergies will be recruited and seen both in and out of allergy season, and 10 healthy controls. Nasal epithelial lining fluid (NELF,) collected by placing small filter papers into the nostrils, blood for analysis and a cold/flu swab will be collected at each study visit.

DETAILED DESCRIPTION:
This is an observational study of adults with and without seasonal allergic rhinitis (AR). Fifty volunteers; 40 with a history of seasonal allergic rhinitis and 10 without a history of allergic rhinitis will be recruited for this study. After screening for eligibility and undergoing informed consent a focused medical history, medication review, and physical exam by the study physician will be performed. An allergic rhinitis questionnaire will be completed by the participant. This will be followed by allergy skin prick testing to a panel of common aeroallergens, collection of NELF samples, a nasal swab and venipuncture. For the non-allergic participants, this will conclude participation in the study. Participants with seasonal allergic rhinitis who completed the first study visit outside of the participant's typical allergy season will return for the second study visit during allergy season, and vice versa for participants presenting for the first study visit during allergy season. For example, a participant with a history of symptomatic allergic rhinitis triggered by tree pollen would attend one study visit during tree pollen season (March-May) and a second study visit outside of allergy season while asymptomatic, a least one month from the first study visit. Participants who suffer from grass pollen allergies would attend the "in-season" study visit during the months of June-August, and participants suffering from weed pollen allergies would attend the "in-season" study visit during the months of September-November. Participants who suffer from allergic rhinitis symptoms related to trees and weeds, but not grass, would attend the "in-season" visit either during March-May or during September-November. For those same participants, the "off-season" visit would occur either during June-August or during December-February.

For each outcome measure, measurements obtained from allergic rhinitics during allergy season and measurements obtained outside of allergy season will be compared. Measurements from samples taken from allergic rhinitics during and outside of allergy season will also be compared with non-allergic sample measurements.

ELIGIBILITY:
Inclusion Criteria:

(Allergic Rhinitics):

* Non-smoking males and females aged 18-70 years, inclusive
* History of Seasonal Allergic Rhinitis defined by:

Sensitization to at least one seasonal aeroallergen via skin prick testing (wheal =3 mm than negative control), AND History of physician-diagnosed seasonal allergic rhinitis, OR Symptoms consistent with seasonal allergic rhinitis, such as runny nose, nasal congestion, sneezing, or nasal pruritis.

* Have lived in the South Atlantic region (Virginia, North and South Carolina, Georgia, Alabama, Florida) for at least 1 year prior to study entry.
* Willing to undergo written informed consent indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Willing and able to comply with scheduled visits, nasal sample collection, and other study procedures.

(Non-allergic):

* Non-smoking males and females aged 18-70 years, inclusive
* No history of physician-diagnosed allergic rhinitis and no history of seasonal runny nose,nasal congestion, sneezing or nasal pruritis.
* Negative results to a panel of aeroallergens via skin prick testing
* Willingness to undergo written informed consent indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Willing and able to comply with scheduled visits, nasal sample collection, and other study procedures.

Exclusion Criteria:

* Symptomatic perennial AR (for example, allergy to dust mite or pet dander causing year-round symptoms)
* Use of immunosuppressive medications such as daily systemic corticosteroids; in addition, participants who have used systemic corticosteroids in the past 3 months will not be enrolled
* Use of other medications or supplements that may interfere with interpretation of outcomes
* Presence of other diagnoses such as non-allergic rhinitis, chronic sinusitis, etc. that in the opinion of the study investigator or medically qualified designee may affect interpretation of the data or subjects' ability to safely participate in the study.
* A subject who is an employee of the investigational site and either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK employee directly involved in the conduct of the study or a member of their immediate family
* A subject who has received treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer)
* A subject who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A subject with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the subject inappropriate for entry into this study
* A subject who is pregnant or intending to become pregnant over the duration of the study
* A subject who is breastfeeding
* Use of tobacco or nicotine products, including electronic cigarettes. A subject who, in the opinion of the investigator or medically qualified designee, should not participate in the study
* Subjects diagnosed with autoimmune diseases
* Subjects with an upper respiratory tract infection within the previous 4 weeks
* Subjects with known nasal polyps
* Subjects with known history of HIV or hepatitis virus
* A subject who has previously been enrolled in this study
* A subject whose gender identity is different from their birth-assigned sex.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the general population, including UNC students and employees, individuals who have participated in previous research studies, and other healthy adults living in the southeastern United States and willing and able.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Eosinophilic Cationic Protein (ECP) in Nasal Epithelial Lining Fluid (NELF) in ng/mL | Up to 15 months
  NELF will be collected from volunteers with a history of seasonal allergic rhinitis. ECP concentration in NELF (ng/mL) will be compared between samples obtained during symptomatic periods (during their relevant allergy season) vs those obtained during asymptomatic periods
Immunoglobulin E (IgE) in NELF in kU/L | Up to15 months
  NELF will be collected from volunteers with a history of seasonal allergic rhinitis. IgE concentration in NELF (ku/L) will be compared between samples obtained during symptomatic periods (during their relevant allergy season) vs those obtained during asymptomatic periods

SECONDARY OUTCOMES:
Respiratory Virus Detection in Nasopharyngeal Swabs | Up to 15 months
  Nasopharyngeal swabs will be performed on volunteers with a history of seasonal allergic rhinitis during symptomatic periods (during their relevant allergy season) and during asymptomatic periods. The percentage of samples containing detectable respiratory virus by Polymerase Chain Reaction (PCR) analysis will be calculated.
Ratio of NELF IgE (kU/L) to Peripheral blood IgE (kU/L) | Up to 15 months
  NELF samples and peripheral blood samples will be obtained at Visit 1. The ratio of IgE in NELF to IgE in peripheral blood will be calculated.
Tryptase in NELF in ng/mL | Up to 15 months
  NELF will be collected from volunteers with a history of seasonal allergic rhinitis. Tryptase concentration in NELF (ng/mL) will be compared between samples obtained during symptomatic periods (during their relevant allergy season) vs those obtained during asymptomatic periods
Inflammatory Cytokines in NELF in pg/mL | Up to 15 months
  NELF will be collected from volunteers with a history of seasonal allergic rhinitis. Inflammatory cytokines in NELF (pg/mL) will be compared between samples obtained during symptomatic periods (during their relevant allergy season) vs those obtained during asymptomatic periods

CONTACTS AND LOCATIONS:
Overall Officials: Neil Alexis, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: 9-36 months following publication

REFERENCES:
- [Background] Gauvreau GM, El-Gammal AI, O'Byrne PM. Allergen-induced airway responses. Eur Respir J. 2015 Sep;46(3):819-31. doi: 10.1183/13993003.00536-2015. Epub 2015 Jul 23. PMID 26206871
- [Background] Arvidsson MB, Lowhagen O, Rak S. Early and late phase asthmatic response in lower airways of cat-allergic asthmatic patients--a comparison between experimental and environmental allergen challenge. Allergy. 2007 May;62(5):488-94. doi: 10.1111/j.1398-9995.2007.01278.x. PMID 17441789
- [Background] Sicherer SH, Wood RA, Eggleston PA. Determinants of airway responses to cat allergen: comparison of environmental challenge to quantitative nasal and bronchial allergen challenge. J Allergy Clin Immunol. 1997 Jun;99(6 Pt 1):798-805. doi: 10.1016/s0091-6749(97)80014-0. PMID 9215248
- [Background] Wenzel S, Wilbraham D, Fuller R, Getz EB, Longphre M. Effect of an interleukin-4 variant on late phase asthmatic response to allergen challenge in asthmatic patients: results of two phase 2a studies. Lancet. 2007 Oct 20;370(9596):1422-31. doi: 10.1016/S0140-6736(07)61600-6. PMID 17950857
- [Background] Deschildre A, Pichavant M, Engelmann I, Langlois C, Drumez E, Pouessel G, Boileau S, Romero-Cubero D, Decleyre-Badiu I, Dewilde A, Hober D, Neve V, Thumerelle C, Lejeune S, Mordacq C, Gosset P. Virus-triggered exacerbation in allergic asthmatic children: neutrophilic airway inflammation and alteration of virus sensors characterize a subgroup of patients. Respir Res. 2017 Nov 14;18(1):191. doi: 10.1186/s12931-017-0672-0. PMID 29137638
- [Background] Kantor DB, Stenquist N, McDonald MC, Schultz BJ, Hauptman M, Smallwood CD, Nelson KA, Perzanowski MS, Matsui EC, Phipatanakul W, Hirschhorn JN. Rhinovirus and serum IgE are associated with acute asthma exacerbation severity in children. J Allergy Clin Immunol. 2016 Nov;138(5):1467-1471.e9. doi: 10.1016/j.jaci.2016.04.044. Epub 2016 Jun 15. No abstract available. PMID 27474123
- [Background] Jaovisidha P, Peeples ME, Brees AA, Carpenter LR, Moy JN. Respiratory syncytial virus stimulates neutrophil degranulation and chemokine release. J Immunol. 1999 Sep 1;163(5):2816-20. PMID 10453026
- [Background] Rebuli ME, Speen AM, Clapp PW, Jaspers I. Novel applications for a noninvasive sampling method of the nasal mucosa. Am J Physiol Lung Cell Mol Physiol. 2017 Feb 1;312(2):L288-L296. doi: 10.1152/ajplung.00476.2016. Epub 2016 Dec 23. PMID 28011618
- [Background] Kaulbach HC, White MV, Igarashi Y, Hahn BK, Kaliner MA. Estimation of nasal epithelial lining fluid using urea as a marker. J Allergy Clin Immunol. 1993 Sep;92(3):457-65. doi: 10.1016/0091-6749(93)90125-y. PMID 8360397
- [Background] Southworth T, Pattwell C, Khan N, Mowbray SF, Strieter RM, Erpenbeck VJ, Singh D. Increased type 2 inflammation post rhinovirus infection in patients with moderate asthma. Cytokine. 2020 Jan;125:154857. doi: 10.1016/j.cyto.2019.154857. Epub 2019 Sep 23. PMID 31557636
- See also: Allergies and Hay Fever U.S. Data — https://www.cdc.gov/nchs/fastats/allergies.htm